CLINICAL TRIAL: NCT04327752
Title: Cutaneous Adverse Effects Occurring in Children Under Biological Therapy Given for Chronic Inflammatory Diseases
Brief Title: Skin Adverse Reactions Occuring in Children Treated by Biotherapy for Chronic Inflammatory Disease
Acronym: MDEBMIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0048
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Biotherapy; Chronic Inflammatory Disease; Allergic Skin Reaction; Pediatric Disorder; Dermatologic Complication; Gastrointestinal Disease; Ophthalmology; Rheumatology
Keywords: Biotherapy; Chronic Inflammatory Disease; skin adverse event; paradoxical reaction; cutaneous manifestation; pediatry; dermatology; gastro-enterology; ophthalmology; rheumatology
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dermatological consultation — Dermatological consultation will be done on every children treated by biotherapy for chronic inflammatory disease in the Amiens hospital.

SUMMARY:
Biological treatments (BT) are commonly prescribed to treat chronic inflammatory diseases in children. Paradoxical reactions during treatment with a biological agent can be defined as the appearance or exacerbation of a pathological condition that usually responds to this class of drug while treating a patient for another condition. Limited data are available in children treated by BT on cutaneous paradoxical reactions, or any other cutaneous adverse events occurring during treatment. On the contrary, dermatologists tend to see and manage increasing numbers of cutaneous adverse events, including paradoxical reactions. The aim of this project is to describe the incidence of cutaneous adverse events, including cutaneous paradoxical reactions, occurring in the pediatric population, during a treatment by BT given for a chronic inflammatory disease.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years old
* Children treated by biotherapy among : Adalimumab, Golimumab, Infliximab, Ustekinumab, Etanercept, Tocilizumab, Canakinumab, Anakinra, Abatacept.
* Children treated for a chronic inflammatory disease (rheumatologic, gastro-enterologic, dermatologic and ophthalmologic)
* Children treated in the CHU of Amiens
* Parental consent signed

Exclusion Criteria:

* Age > 18 ans

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * For the children already under biological therapy for an inflammatory chronic disease : they will benefit of one dermatologic consultation at any time of their treatment. Other consultations can be asked by the patient or by his parents if any skin manifestation appears beside the planned date of the consultation.
  * For the children who are going to be treated by a biological therapy : they will benefit of one dermatologic consultation BEFORE the onset of the biological therapy, and on other one at 4 months afetr the beginning of the treatment. Other consultations can be asked by the patient or his parents if any skin manifestation appears beside the planned dates of both consultations.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Variation of the incidence of cutaneous adverse events under biological therapy | up to 8 months
  Determine the variation of the incidence of any skin manifestation under biological therapy, including Paradoxical Reaction (psoriasis, eczema, hidradenitis suppurativa …), non-paradoxical inflammatory reaction, infection, neoplasia, hair and nail manifestation, xerosis.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No